CLINICAL TRIAL: NCT00367237
Title: A Randomized, Multicenter, International, Open-label Study of Infliximab Plus Methotrexate Versus Methotrexate (MTX) Alone for the Treatment of MTX naïve Subjects With Active Psoriatic Arthritis
Brief Title: Remicade Study in Psoriatic Arthritis Patients Of Methotrexate-Naïve Disease (RESPOND) (Study P04422)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Integrated Therapeutics Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04422; EUDRACT #: 2005-002189-12
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Infliximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab + methotrexate (IFX + MTX) (Experimental): Remicade (infliximab [IFX]) 5 mg/kg infusions at Weeks 0, 2, 6, 14 and oral methotrexate (MTX) 15 mg/week
  Interventions: Drug: Infliximab + methotrexate (IFX + MTX)
- Methotrexate (MTX) (Active Comparator): Oral methotrexate (MTX) 15 mg/week
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Infliximab + methotrexate (IFX + MTX) — Infliximab 5 mg/kg infusion at Weeks 0, 2, 6, 14 and oral methotrexate 15 mg/week for 16 weeks. Methotrexate dose can be increased to 20 mg/week at week 6.
  Other Names: Group 1, Remicade + MTX
  Arms: Infliximab + methotrexate (IFX + MTX)
Drug: Methotrexate (MTX) — Oral methotrexate 15 mg/week for 15 weeks. Dose can be increased to 20 mg/week at Week 6.
  Other Names: Group 2, MTX
  Arms: Methotrexate (MTX)

SUMMARY:
This study is undertaken to compare the efficacy and onset of action of infliximab plus methotrexate (IFX + MTX) versus methotrexate alone (MTX) in methotrexate naïve active psoriatic arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject must meet ALL of the criteria listed below for entry into the study:
* Subject must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subject aged 18 years or more, of either sex and any race
* Diagnosis of Psoriatic Arthritis with peripheral polyarticular involvement. Patients will have at least one of the following:

  * Distal Interphalangeal Joints (DIP) involvement
  * polyarticular arthritis, absence of rheumatoid nodules and presence of psoriasis
  * arthritis mutilans
  * asymmetric peripheral arthritis
* Negative rheumatoid factor
* The disease should have been diagnosed at least 3 months prior to screening.
* Active disease at the time of screening and prior to receiving the baseline study medication(s) as defined by:

  * 5 or more swollen joints and
  * 5 or more tender joints
  * and one out of the following three categories:

    * Erythrocyte Sedimentation Rate (ESR) >= 28 mm/h
    * C-reactive protein (CRP) >= 15 mg/l
    * Morning stiffness >= 45 min
* Subjects must confirm that they are practicing adequate contraception: Female subjects of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active during the study) must agree to use a medically accepted method of contraception or be surgically sterilized prior to screening, while receiving protocol-specified medication, and for 6 months after stopping the medication. Acceptable methods of contraception include condoms (male and female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), oral or injectable hormonal contraceptive, and surgical sterilization (e.g., hysterectomy or tubal ligation).
* Female subjects of childbearing potential must have a negative pregnancy test at Screening.
* Subjects must be eligible for anti-tumor necrosis factor (TNF) treatment according to applicable local guidelines. For all patients chest X-ray and skin test results must be available at baseline.
* If using Nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids other than i.v., i.m. or i.a., the patient must be on a stable dose for four weeks prior screening (maximum dose up to 10mg/day of prednisone or its oral equivalent).
* The screening laboratory tests must beet the following criteria:

  * Hemoglobin >= 10 g/dl providing the low hemoglobin level is not due to other diseases than anemia of chronic inflammation.
  * white blood cell (WBC) >= 3500 / μl
  * Neutrophils >= 1500 / μl
  * Platelets >= 100 000/ μl
  * Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, and gamma-glutamyltransferase <= 1.5 x upper limit of normal
  * Total bilirubin <= 1 x upper limit of normal
  * Serum creatinine <= 1.5 mg/dl
* Patient must be able to adhere to the study visit schedule and other protocol requirements and must have given informed consent prior to any screening procedures.

Exclusion Criteria:

* The subject will be excluded from entry into the study if ANY of the criteria listed below are met:
* Subject is a female who is pregnant, intends to become pregnant during the study (or within 6 months after study completion), or nursing.
* Patients with other inflammatory diseases that might interfere with the evaluation of the psoriatic arthritis.
* Previous treatment with Infliximab.
* Subjects who have previously received MTX or have not discontinued their other DMARD therapy (i.e., sulfasalazine, hydroxychloroquine, leflunomide).
* Patients with fibromyalgia syndrome.
* Use of cyclosporine or tacrolimus within 4 weeks prior to screening. Use of IM, IV, or IA corticosteroids within 4 weeks prior to screening.
* Treatment with any investigational drug within 3 months prior to screening.
* Previous treatment with a monoclonal antibody or a fusion protein.
* A history of known allergy to murine proteins.
* History of infected joint prosthesis within the previous 5 years.
* Chronic infections.
* History of active tuberculosis requiring treatment within previous 3 years or history of opportunistic infections within 2 months, uncontrolled active infection or documented HIV infection. Also excluded are patients with evidence of latent tuberculosis and patients with old tuberculosis without documented adequate therapy, if they will not be treated according to local tuberculosis (TB) guidelines.
* Subject has any clinically significant deviation from normal in the physical examination, chest X-ray, or electrocardiogram (ECG) that, in the investigator's judgment, may interfere with the study evaluation or affect subject safety.
* Current signs or symptoms of other severe uncontrolled diseases, which in the investigators opinion would put the patient at an unacceptable risk.
* History of lymphoproliferative disease, any current malignancies or history of malignancy within 5 years other than successfully treated basal cell carcinoma or squamous cell carcinoma of the skin.
* Subject is part of the staff or a family member of the staff personnel directly involved with this study.
* History of drug abuse.
* Subjects who are participating in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Baranauskaite A, Raffayova H, Kungurov NV, Kubanova A, Venalis A, Helmle L, Srinivasan S, Nasonov E, Vastesaeger N; RESPOND investigators. Infliximab plus methotrexate is superior to methotrexate alone in the treatment of psoriatic arthritis in methotrexate-naive patients: the RESPOND study. Ann Rheum Dis. 2012 Apr;71(4):541-8. doi: 10.1136/ard.2011.152223. Epub 2011 Oct 12. PMID 21994233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 subjects (57 infliximab (IFX) + MTX and 58 MTX), but only 110 subjects (56 and 54) were considered intent to treat (ITT). Furthermore, 99 subjects (51 + 48) were in a treatment group at Week 16 for Primary Endpoint evaluation.
Period: Overall Study
Arm/Group | Infliximab + Methotrexate (IFX + MTX) | Methotrexate (MTX)
Started | 57 (Number of subjects randomized) | 58 (Number of subjects randomized)
Completed | 47 | 47
Not Completed | 10 | 11
Not completed — Adverse Event | 7 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Protocol Violation | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab + Methotrexate (IFX + MTX) | Methotrexate (MTX) | Total
Number analyzed (Participants) | 56 | 54 | 110
Age, Continuous [Mean (Full Range); unit: years] — ITT population
  years | 40.1 [20 to 65] | 42.3 [21 to 65] | 41.2 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 21 | 50
  Male | 27 | 33 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving ACR20 (at Least 20% Improvement in American College of Rheumatology Criteria From Baseline) at Week 16
Description: >=20% improvement in swollen and tender joint count AND >=20% improvement in 3 of the following: visual analog scale (VAS) assessment of pain; subject VAS global assessment of disease activity; evaluator VAS global assessment of disease activity; Health Assessment Questionnaire (HAQ) disability index; C-Reactive Protein (CRP) level.
Time Frame: between baseline and week 16
Population: Number of subjects from Intent-to-Treat population in each arm at Week 16
Measure: Number; unit: participants
Arm/Group | Infliximab + Methotrexate (IFX + MTX) | Methotrexate (MTX)
Number analyzed (Participants) | 51 | 48
participants | 44 | 32
Statistical Analysis 1: Comparison: Infliximab + Methotrexate (IFX + MTX) vs Methotrexate (MTX); Test type: Superiority or Other; p = 0.0210, Chi-squared — Comparison of treatments (IFX + MTX versus MTX); Difference in percentages of respondents = 19.61, 95% CI [3.27 to 35.95] — Difference in percentages of respondents is (percentage of respondents in IFX+MTX group minus percentage of respondents in MTX group)
Statistical Analysis 2: Comparison: Infliximab + Methotrexate (IFX + MTX); Test type: Superiority or Other; Proportion of Responders = 0.863
Statistical Analysis 3: Comparison: Methotrexate (MTX); Test type: Superiority or Other; Proportion of Responders = 0.667

2. Secondary Outcome: Proportion of Subjects Achieving ACR50, ACR70, and PASI75 if Applicable
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: between baseline and week 16
Reporting Status: Not Posted

3. Secondary Outcome: Change in Disease Activity Score, Each of the ACR20 Domains, Dactylitis, Enthesitis, Fatigue and Duration of Morning Stiffness, Erythrocyte Sedimentation Rate, and Disability Index of the Health Assessment Questionnaire (HAQ)
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: between baseline and week 16
Reporting Status: Not Posted

4. Secondary Outcome: Adverse Events
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: between baseline and week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety analyses included all subjects who received at least 1 dose of study medication
  Subjects were questioned and/or examined by the investigator for evidence of adverse events. The questioning of subjects with regard to the possible occurrence of adverse events were to be generalized such as, "How have you been feeling since your last visit?"
Arm/Group | Infliximab + Methotrexate (IFX + MTX) | Methotrexate (MTX)
Serious Adverse Events (participants affected / at risk) | 2/57 | 0/54
Other Adverse Events (participants affected / at risk) | 12/57 | 10/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab + Methotrexate (IFX + MTX) (N=57) | Methotrexate (MTX) (N=54)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab + Methotrexate (IFX + MTX) (N=57) | Methotrexate (MTX) (N=54)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 6 (6) | 5 (5)
Blood Bilirubin Increased (Investigations) | 2 (2) | 3 (3)
Transaminases Increased (Investigations) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator must provide 30 days written notice to sponsor prior to submission for publication/presentation, so that sponsor can review the material(s). If the parties disagree concerning the appropriateness of the material for publication, the investigator must meet with sponsor prior to publication/presentation, in order to make good faith efforts to discuss and resolve any disagreements.